CLINICAL TRIAL: NCT06017011
Title: Clinico-Radiological Characterisation for Remission of Acute Charcot-Neuroarthropathy of Foot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: C- PRIME Study
Record Dates: First submitted 2023-03-19; First posted 2023-08-30 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Acute Charcot Neuroarthropathy
Keywords: Charcot neuroarthropathy; F18 Fluoride PET scan; MRI of the Foot; RANKL; Osteoprotegerin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for the estimation of free soluble RANKL and Osteoprotegerin levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute charcot neuroarthropathy or Acute on Chronic charcot neuroarthropathy: Patients diagnosed with Acute charcot neuroarthropathy or Acute on Chronic charcot neuroarthropathy will be put on Total contact cast and followed till clinical remission and then after that till 6 months post clinical remission.
  Interventions: Other: Total contact cast

INTERVENTIONS:
Other: Total contact cast — Total contact cast will be put on the patient at the diagnosis of Acute charcot neuroarthropathy and the patient will be followed till clinical remission and after that till 6months post clinical remission. F18 Fluoride PET scan and MRI of the foot with DWI and ADC sequence to be done at baseline, Clinical remission, 3months post clinical remission and 6months post clinical remission to quantitate the process of remission.

SUMMARY:
Charcot's neuro-arthropathy is a condition which is generally prevalent among the diabetic patients. Acute charcot's neuro-arthropathy is characterized by signs of inflammation, hot, red swelling around the involved joint along with a temperature difference of greater than 2 degree centigrade between the two feet. This is often misdiagnosed as cellulitis, sprains or deep vein thrombosis. The diagnosis of this condition is mainly made clinically and aided by x-ray of foot, MRI of foot and sometimes by bone scan. The therapy that is accepted unanimously is putting on a total contact cast. The duration of this therapy depends on the regular temperature monitoring of both the feet. When the temperature difference between the two feet comes down to less than 2 degree centigrade, then it is defined as clinical remission and the offloading of the foot is stopped. There are other modalities that have been tried for the treatment of acute charcot's neuro-arthropathy with medications like methyl prednisolone, bisphosphonates and the effects of medical management of acute charcot's neuro-arthropathy was a mixed one with no definite recommendation regarding use of medical management in this condition. If the patients are denied these treatment then there is progression of the disease process and can lead to the development of chronic changes in the form of fractures, dislocation, gangrene, foot ulcers and ultimately amputation. The end point of the treatment with total contact cast is taken as the decrease in the temperature difference of less than 2 degree centigrade between the two feet. This point is regarded as the point of clinical remission in cases of acute charcot's neuro-arthropathy. But there has been instances where there have been 12-33% of recurrences when this clinical remission has been used as a criteria for discontinuation of offloading. With time, there has been evolution in the imaging of charcot's neuro-arthropathy. There has been advent of MRI and MRS of the foot for monitoring of acute charcot's neuro-arthropathy remission which is the most sensitive technique for the recognition of early bony changes in charcot neuro-arthropathy. PET scan has also been used including bone scan and FDG PET scan, for the evaluation of acute charcot's neuro-arthropathy remission. Even with these modalities the actual remission criteria that would decrease the complication of early offloading as done at the time of clinical remission, is still missing. So here the investigators aim to monitor the process of remission of acute charcot-neuroarthropathy of foot both clinically as well as radiologically with the help of MRI of the foot with diffusion weighted and apparent diffusion coefficient imaging along with a novel PET scan for charcot's neuroarthropathy, that is F18-Fluoride PET scan which will given a quantitative estimation of the process of remission of acute charcot-neuroarthropathy in the form of SUV max. Thus this quantitative value can help to assess the trends of remission in acute charcot neuroarthropathy of foot.

DETAILED DESCRIPTION:
Charcot's neuro-arthropathy is a condition which is generally prevalent among the diabetic patient. It is a condition which primarily affects the bones and the joints. The presentation of charcot's neuro-arthropathy can be an acute or a chronic type depending upon the temperature difference between the two feet i.e. greater than 2 degree centigrade. Acute charcot's neuro-arthropathy presents with signs of redness, swelling and raised temperature of the involved area. The condition if not detected in the acute condition leads to chronic changes in the joints which leads to joint dislocation, fractures and development of rocker-bottom foot and also can lead to a state where amputation of the affected foot is needed. Acute charcot's neuro-arthropathy is characterized by signs of inflammation, hot, red swelling around the involved joint. This is often misdiagnosed as cellulitis, sprains or deep vein thrombosis. The diagnosis of this condition is mainly made clinically and aided by x-ray of foot, MRI of foot and sometimes by bone scan. The therapy that is accepted unanimously is putting on a total contact cast. The duration of this therapy depends on the regular temperature monitoring of both the feet. When the temperature difference between the two feet comes down to less than 2 degree centigrade, then it is defined as clinical remission and the offloading of the foot is stopped. Keeping in mind the effects of RANKL in the pathogenesis of acute Charcot neuro-arthropathy, Zoledronic acid was used as a treatment modality for acute charcot neuro-arthropathy. But it showed that it was inferior to the application of total contact cast. There have been trials were methylprednisolone combined with total contact cast have been used for treatment and the outcome has been compared with the use of zoledronate in patients on total contact cast. It had shown that zoledronate with total contact cast had an improvement of bone mineral density and on the other hand there was a decrease with steroids. Overall the effects of medical management of acute charcot's neuro-arthropathy was a mixed one with no definite recommendation regarding use of medical management in this condition. So total contact cast is the gold standard for the management of acute charcot's neuro-arthropathy. It has led to the healing of ulcers to the range of 75% in cases of acute charcot's neuro-arthropathy. If the patients are denied these treatment then there is progression of the disease process and can lead to the development of chronic changes in the form of fractures, dislocation, gangrene, foot ulcers and ultimately amputation.

The end point of the treatment with total contact cast is taken as the decrease in the temperature difference of less than 2 degree centigrade between the two feet. This point is regarded as the point of clinical remission in cases of acute charcot's neuro-arthropathy. But there has been instances where there have been 12-33% of recurrences when this clinical remission has been used as a criteria for discontinuation of offloading.

There has been advent of MRI and MRS of the foot for monitoring of acute charcot's neuro-arthropathy remission which is the most sensitive technique for the recognition of early bony changes in charcot neuro-arthropathy. PET scan has also been used including bone scan and FDG PET scan, for the evaluation of acute charcot's neuro-arthropathy remission. These modalities have been evaluated to test the actual remission of acute charcot's neuro-arthropathy. Even with these modalities the actual remission criteria that would decrease the complication of early offloading as done at the time of clinical remission, is still missing.

There is no quantitative method available to monitor the process of remission of acute charcot-neuroarthropathy and accurately label the remission.

The pathophysiology of acute charcot neuro-arthropathy has two main postulates. One is the neurovascular theory in which it is thought to have nerve damage and it leads to increased local vascularity which leads to activation of increased osteoclastic activity with development of secondary osteopenia, fractures and deformity. The other theory is the more accepted one and has attracted a lot of recent research around it. This involves the neuro-traumatic theory where due to the presence of neuropathy in these diabetic patients, they are not able to realize the microtrauma that they sustain. This leads to the development of a state of inflammation resulting in the raised levels of raised IL6 and TNFalpha. There is also activation of the RANKL and OPG pathways leading to bone destruction. This highlights the importance of RANKL in the pathogenesis of acute charcot neuro-arthropathy.

Earlier bone scan, MR Spectroscopy, FDG PET scan has been used to evaluate quantitatively the process of remission of acute charcot-neuroarthropathy. Here we try to quantitate the process of remission of acute charcot neuroarthropathy by using F18- Fluoride PET scan of the foot along with MRI of the foot with Diffusion weighted and apparent diffusion coefficient imaging sequences.

F18- Fluoride PET scan is a modality that is highly sensitive for bone related pathology. It gets attached to area where there is increased osteoblastic activity. The mechanism of skeletal uptake of 18F-NaF is based on ion exchange, which is similar to that of 99mTc-MDP. Bone has a strong architecture and it is due to a crystalline matrix of calcium and phosphate known as hydroxyapatite, which is composed of many different positive and negative ions. 18F ions is exchanged with hydroxyl ions (OH-) on the surface of the hydroxyapatite to form fluoroapatite. The sensitivity of F18 Fluoride PET Scan is also higher than the F18 FDG PET scan as well as bone scan for bone related pathologies. Pathologically altered osteoblastic activity is most efficiently taken up by 18F-NaF-PET, which detects incident photons that results from positron emission of radioactive fluoride ions that have become incorporated into the hydroxyapatite surface of newly formed bone.

It has still not been used in monitoring of remission of acute charcot neuro-arthropathy but as this gives a quantitative value in the form of SUV, so it can be used in the monitoring of acute charcot neuro-arthropathy remission.

MRI of the Foot with Diffusion Weighted Imaging (DWI) sequence in the MRI is used to see if there is any restriction of the brownian motion. It helps to detect conditions where there is restriction of the brownian motion like infection. DWI sequence also has an advantage in that it helps to differentiate osteomyelitis from acute charcot-neuro-arthropathy. Apparent Diffusion Coefficient (ADC) sequence can give a semi-quantitative value by plotting the graph from the obtained imaging of the foot and thus it may help in the monitoring of remission.

It has been postulated that RANKL plays a very pivotal role in the process of development of acute charcot neuro-arthropathy. The increased levels of RANKL leads to the activation of the osteoclastic activity and there is extensive destruction of the joints seen. RANKL has been used for studying the process of remission in acute charcot neuro-arthropathy. It has been studied that during the follow up of two years in the patients of acute charcot neuro-arthropathy after the application of total contact cast, there was significant decrease in the levels and it had come down to comparable values with the healthy controls.

Osteoprotegerin is another biomarker that has attracted attention for research. This is generally involved in the inhibition of osteoclastic activity. So in areas where there is increase in the osteoclastic activity and elevation of the RANKL, there is also similar elevation of the OPG levels as well as the osteoclastic and the osteoblastic activities which go hand in hand.

So here the investigators want to use these quantitative imaging tools and biochemical markers to assess the trends of remission in acute charcot neuroarthropathy and compare it with clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Diabetes,

  1. Diagnosed both clinically as well as radiologically to be having unilateral acute charcot neuro-arthropathy.
  2. Irrespective of age, glycemic status, CKD staging.

Exclusion Criteria:

-1) The patients who are contraindicated for MRI like metallic implants, Pace maker in situ.

2) Active infected foot ulcers 3) Osteomyelitis 4) Patients on drugs altering bone metabolism like bisphosphonates, teriparatide, Denosumab in the past 2 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Diabetes diagnosed with acute charcot neuroarthropathy or acute on chronic charcot neuroarthropathy.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax change in F18 Fluoride PET scan | From baseline till 6 months post clinical remission
  To assess the quantitative change in SUVmax in F18- Fluoride PET of the foot from diagnosis to 6months post clinical remission and calculate the cutoff/ Delta (change in SUVmax) in comparison to clinical remission in acute charcot neuro-arthropathy.

SECONDARY OUTCOMES:
ADC values of the MRI Foot with DWI and ADC | From baseline to 6 months post clinical remission
  To assess the trends of ADC values of the MRI Foot with DWI and ADC sequences from baseline to 6months post clinical remission in acute charcot-neuroarthropathy
RANKL and Osteoprotegerin | From baseline to 6 months post clinical remission
  To assess the role of biomarkers and imaging in monitoring the remission of acute charcot neuro-arthropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Ashu Rastogi, MD, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No